CLINICAL TRIAL: NCT01905007
Title: "Test-No Test" Implantable Cardioverter Defibrillator Pilot Study (TNT-ICD)
Brief Title: Study of Defibrillation Testing In Patients Undergoing Initial ICD Implantation
Acronym: TNT-ICD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Collaborators: Medtronic (Industry); University of Washington (Other)
Responsible Party: Principal Investigator, Andrea M. Russo, MD, Professor of Medicine, Director of Electrophysiology & Arrhythmia Services, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUH-09-087
Record Dates: First submitted 2012-02-24; First posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Ventricular Arrhythmias
Keywords: Implantable cardioverter defibrillator; Defibrillation threshold testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Defibrillation testing (Active Comparator): Defibrillation testing at initial ICD implantation
  Interventions: Device: Defibrillation testing
- No defibrillation testing (No Intervention): No defibrillation testing at initial ICD implantation

INTERVENTIONS:
Device: Defibrillation testing — Defibrillation testing at initial ICD implantation
  Other Names: Medtronic implantable cardioverter defibrillator
  Arms: Defibrillation testing

SUMMARY:
The primary objective of this study is to compare the composite outcome of total mortality and operative complications in patients who do not undergo defibrillation testing to those who do undergo defibrillation testing at the time of initial ICD implantation.

DETAILED DESCRIPTION:
Implantable cardioverter-defibrillators (ICDs) are the most effective treatment for the primary and secondary prevention of sudden cardiac death (SCD). At the time of ICD implantation, ventricular fibrillation (VF) is typically induced to demonstrate effective arrhythmia termination by the implanted device. Although defibrillation threshold (DFT) testing with induction of VF at time of ICD insertion is currently considered the "standard of care," and instructions for usage of devices approved by the Food and Drug Administration (FDA) include labeling with DFT testing, the value of defibrillation testing with modern-day devices has been questioned. Defibrillation testing can be associated with serious complications and may add to the cost of the procedure.

It is hypothesized that patients who do not undergo defibrillation testing will have outcomes similar to those who do undergo defibrillation testing at the time of initial implantation. This pilot study is being performed to determine the feasibility of performing a larger, multi-center clinical trial with longer follow-up to investigate whether or not defibrillation testing will have any impact on overall mortality, implant complications, or long-term first shock efficacy during clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Initial ICD implantation (single, dual, or CRT) for a standard Class I or Class II indication according to the ACC/AHA/HRS practice guidelines
* Anticipated life expectancy >6 months

Exclusion Criteria:

* Contraindications to defibrillation testing as determined by the managing physician*
* ICD replacement implants
* Right-sided pectoral implants
* Abdominal implants
* Chronic oral amiodarone therapy (for >6 weeks and continued need for amiodarone)
* Inability to give informed consent

  * Contraindications to defibrillation testing include the following: hemodynamic instability, LA thrombus, atrial fibrillation without adequate anticoagulation, LV thrombus, recent CVA or TIA, severe unrevascularized coronary artery disease or unstable angina, severe aortic stenosis, inotropic dependence, patient refusal, other patient-specific medical conditions that are deemed as contraindications, as determined by the implanting physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Composite all-cause mortality and operative complications | Procedure-related complications will be defined as those occurring within 90 days post-implantation and mortality will be measured at 2 year follow-up
  The composite endpoint of implant complications and mortality rates will be compared in the DFT vs. no DFT groups.

SECONDARY OUTCOMES:
1st shock efficacy for clinical occurrence of ventricular tachycardia (VT)/VF | 2 years
  The efficacy of 1st shock therapy for VT/VF will be compared between the DFT and no DFT groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M. Russo, MD, Principal Investigator — The Cooper Health System
Locations (2):
- United States (2):
  - Cooper University Hospital, Camden, New Jersey
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Russo AM, Sauer W, Gerstenfeld EP, Hsia HH, Lin D, Cooper JM, Dixit S, Verdino RJ, Nayak HM, Callans DJ, Patel V, Marchlinski FE. Defibrillation threshold testing: is it really necessary at the time of implantable cardioverter-defibrillator insertion? Heart Rhythm. 2005 May;2(5):456-61. doi: 10.1016/j.hrthm.2005.01.015. PMID 15840466
- [Background] Swerdlow CD, Russo AM, Degroot PJ. The dilemma of ICD implant testing. Pacing Clin Electrophysiol. 2007 May;30(5):675-700. doi: 10.1111/j.1540-8159.2007.00730.x. PMID 17461879
- [Background] Mainigi SK, Cooper JM, Russo AM, Nayak HM, Lin D, Dixit S, Gerstenfeld EP, Hsia HH, Callans DJ, Marchlinski FE, Verdino RJ. Elevated defibrillation thresholds in patients undergoing biventricular defibrillator implantation: incidence and predictors. Heart Rhythm. 2006 Sep;3(9):1010-6. doi: 10.1016/j.hrthm.2006.05.028. Epub 2006 Jun 15. PMID 16945792
- [Background] Blatt JA, Poole JE, Johnson GW, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Anderson J, Chung K, Wong WS, Mark DB, Lee KL, Bardy GH; SCD-HeFT Investigators. No benefit from defibrillation threshold testing in the SCD-HeFT (Sudden Cardiac Death in Heart Failure Trial). J Am Coll Cardiol. 2008 Aug 12;52(7):551-6. doi: 10.1016/j.jacc.2008.04.051. PMID 18687249
- [Background] Birnie D, Tung S, Simpson C, Crystal E, Exner D, Ayala Paredes FA, Krahn A, Parkash R, Khaykin Y, Philippon F, Guerra P, Kimber S, Cameron D, Healey JS. Complications associated with defibrillation threshold testing: the Canadian experience. Heart Rhythm. 2008 Mar;5(3):387-90. doi: 10.1016/j.hrthm.2007.11.018. Epub 2007 Nov 28. PMID 18243813
- [Background] Pires LA, Johnson KM. Intraoperative testing of the implantable cardioverter-defibrillator: how much is enough? J Cardiovasc Electrophysiol. 2006 Feb;17(2):140-5. doi: 10.1111/j.1540-8167.2005.00294.x. PMID 16533250